CLINICAL TRIAL: NCT05124353
Title: Evaluation of the Effect of Early Administration of Neuroprotective Drug (Cerebrolysin) on the Outcome of Patients With Acute Ischemic Stroke Undergoing Endovascular Therapy
Brief Title: Early Administration of Cerebrolysin on the Outcome of Patients With Acute Stroke Undergoing EVT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Klaudyna Kojder, Principal Investigator, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neuroprotective 1/2021
Record Dates: First submitted 2021-06-25; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Stroke, Acute, Ischemic
Keywords: acute.stroke; ischemic stroke; neuroprotection; treatment
MeSH Terms: conditions — Ischemic Stroke | interventions — cerebrolysin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- G1 : Treatment Group (TG)r (Active Comparator): Patients in TG receive neuroprotective drug: standard dose of Cerebrolysin 30ml i.v. in the first 6 hours after first symptoms. After EVT the administration is continued for 10 days.
  Interventions: Drug: Cerebrolysin
- G2 : Control Group (CG) (No Intervention): Patients in CG receive no additional i.v. treatment.

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin 30ml i.v., administrated in first 6 hours after stroke onset and fo 10 day afterwards in Neurology Department or ICU conditions.
  Other Names: neuroprotective treatment
  Arms: G1 : Treatment Group (TG)r

SUMMARY:
Background:

Stroke is the third major cause of death and disability worldwide. It was shown that combining early reperfusion therapy (thrombolysis and/or thrombectomy) with stroke unit care and immediate rehabilitation have beneficial effects on the patient recovery and outcomes. Cerebrolysin that was proven to have s neuroprotective and neurotrophic effects in vitro and in vivo, administered in combination with endovascular therapy (EVT) could have a positive impact on the prognosis and outcome of these patients.

Objectives:

To evaluate the impact of early administration of neuroprotective drug (Cerebrolysin) in patient undergoing EVT on the outcome of patients diagnosed with acute ischemic stroke.

Methods:

100 patients will be recruited to the proposed study according to the inclusion criteria:

Inclusion criteria:

Acute ischemic stroke patients NIHSS>8 Qualification for mechanical thrombectomy, without previous thrombolysis. The patients will be randomized into 2 subgroups: G1(standard dose of Cerebrolysin 30ml), - G2 (No Cerebrolysin).

The patients will be randomized into 2 subgroups: G1(standard dose of Cerebrolysin 30ml), - G2 (No Cerebrolysin). Cerebrolysin will be administered immediately after randomization or at the latest during the EVT procedure and will be continued for 10 days. After the EVT all patients, depending on their clinical condition, will be hospitalized in ICU (intensive care unit) or Neurology Department, where standard treatment and monitoring will be implemented, as well as standard rehabilitation. Outcome assessments will include: the NIH Stroke Scale, modified Rankin Score, pre MRS, IQ code, Geriatric Depression Scales, MoCA. Additionally, the infarct volume of the control CT will be measured. The follow up should be performed on day 7( or discharge), 1 month, 3 months, 6 months. The duration of the study is planned forr: 12 -24 months

DETAILED DESCRIPTION:
Introduction:

Acute ischemic stroke is one of the main leading cause of death and disability in the world. In proposed project we evaluate the impact of the combination of early reperfusion therapy (thrombectomy) with early neuroproptective drug administration on treatment results in patients with acute ischemic stroke. Cerebrolysin, which has been shown to have neuroprotective and neurotrophic effects in vitro and in vivo, when administered early in combination with early endovascular therapy may have a positive effect on the prognosis and treatment outcomes of these patients. The proposed study, is approved by the Pomeranian Medical University Bioethics Committee in Szczecin, Poland, will be also part of the international CERECAP project investigating the co-application of neuroprotective and reperfusion therapies (thrombolysis, thrombectomy) in patients with acute ischemic stroke.

Purpose of the project:

examining the impact of early cerebrolysin supply on the treatment effect in patients with diagnosed acute ischemic stroke, qualified for endovascular treatment in the form of thrombectomy

Hypothesis:

Cerebrolysin in early (up do 6 h) administration with combination of early (up to 6h) endovascular therapy (thrombectomy) is beneficial for the patients with acute ischemic stroke diagnosis.

Material and method 100 patients will be qualified for the proposed project. Study duration: 24 months.

Inclusion criteria for the study diagnosis of acute ischemic stroke qualification for endovascular treatment in the form of thrombectomy

Criteria for exclusion from the study:

Patient qualified for thrombolysis Patients under 18 years of age pregnancy Kidney failure Epilepsy History of allergy to cerebrolysin

Study design:

After prior randomization to the group, patients will be divided into group G1 (cerebrolysin supply) and group G2 (standard treatment, without cerebrolysin supply).

In group G1, cerebrolysin will be administered immediately after qualifying for the study (i.e. up to 6 hours after the onset of symptoms) and continued for the next 10 days at a dose of 30 ml i.v.

Patients from both groups G1 and G2 will undergo thrombectomy treatment, and then, depending on the clinical condition, hospitalized in the Intensive Care Unit or the Department of Neurology with the Stroke Department.

During the hospitalization, the standard and typical care for both departments will be continued.

Treatment results will be assessed using:

NIH, Modified Rankin Scale, preMRS, IQ code, Geriatric Depression Scale and MoCA.

Routine checkups for computed tomography will also undergo analysis for treatment evaluation (e.g. stroke volume). Patients' condition will be assessed after 1, 3 and 6 months.

The results obtained in this way will be statistically analyzed and presented in the form of articles in medical journals.

Expected benefits:

* examination of the influence of early cerebrolysin supply on the treatment effect in patients undergoing thrombectomy after acute ischemic stroke diagnosis
* development of the cerebrolysin supply protocol in patients with acute ischemic stroke diagnosis

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke diagnosis,
* qualification for mechanical thrombectomy, without previous thrombolysis
* age >18

Exclusion Criteria:

* age <18
* pregnancy
* cerebrolysin allergy
* epilepsy
* renal failure
* thrombolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 6 months
  survival rate within first 6 months
NIHSS | day 1
  NIH Stroke Scale
NIHSS | month 3
  NIH Stroke Scale
NIHSS | month 6
  NIH Stroke Scale
Rankin | day 1
  modified Rankin Score
Rankin | month 3
  modified Rankin Score
Rankin | month 6
  modified Rankin Score
pre MRS | day 1
  modified pre Rankin Score
pre MRS | month 3
  modified pre Rankin Score
pre MRS | month 6
  modified pre Rankin Score
IQ code | month 3
  IQ code
IQ code | month 6
  IQ code
Geriatric Depression Scales | month 3
  Geriatric Depression Scales
Geriatric Depression Scales | month 6
  Geriatric Depression Scales
IV | 10 days
  infarct volume of the control CT
modified treatment in cerebral infarction (mTICI score) | 1 month
  measure the reperfusion grade post thrombectomy - radiological imaging

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Jarosz, Principal Investigator — Pomeranian Medical Univerisity
Locations (1):
- Pomeranian Medical University, University Hospital no.1, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: No